CLINICAL TRIAL: NCT05056168
Title: Validation of a Dermatology-Specific Treatment Satisfaction Instrument
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, April Armstrong, Professor, University of Southern California
Other Study IDs: HS-18-00891-AM004
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dermatology-Specific Treatment Satisfaction Instrument — Study subjects will also be administered a dermatology-specific treatment satisfaction questionnaire, as well as other questionnaires including the generic validated Treatment Satisfaction Questionnaire for Medication (TSQM-9) and the validated Dermatology Life Quality Index (DLQI). Study participants will also self-report their disease severity using PGA. Depending on patients' preferred method of interacting with the study team, the investigators will collect their responses to these questionnaires either in-person, over the phone, or electronically via secure research platforms.

SUMMARY:
The primary objective of this study is to validate a dermatology-specific questionnaire that assesses patient satisfaction with their treatments across various inflammatory dermatology diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years)
* Psoriasis patients undergoing some form of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥ 18 years) dermatology patients with psoriasis from LAC+USC and Keck Medical Centers, the Brigham and Women's Hospital, and the Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of a dermatology-specific treatment satisfaction instrument in patients with psoriasis | 8 months
  For this survey study, the investigators will gather descriptive statistics for each item in the questionnaire. The investigators will also measure the following psychometric properties: measurement error, reliability and construct validity, as measured by convergent and known-groups validity

CONTACTS AND LOCATIONS:
Overall Officials: April Armstrong, MD, MPH, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States